CLINICAL TRIAL: NCT03252379
Title: Endoscopic Access Loop With Bilio-enteric Anastomosis: A Prospective Randomized Comparison Between Gastric and Subcutaneous Accesses
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamad Raafat, Assistant lecturer at General surgery department, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RF2017
Record Dates: First submitted 2017-08-12; First posted 2017-08-17 (Actual); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Jaundice, Obstructive
MeSH Terms: conditions — Jaundice, Obstructive

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into three groups according to the surgical procedure performed as follows:
  * Group A: Patients undergoing modified hepaticojejunostomy with gastric access loop
  * Group B: Patients undergoing modified hepaticojejunostomy with subcutaneous access loop
  * Group C: Patients undergoing standard hepaticojejunostomy with no endoscopic access loop
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Patients undergoing modified hepaticojejunostomy with gastric access loop
  Interventions: Procedure: modified hepaticojejunostomy with gastric access loop
- Group B: (Experimental): Patients undergoing modified hepaticojejunostomy with subcutaneous access loop
  Interventions: Procedure: modified hepaticojejunostomy with subcutaneous access loop
- Group C: (Experimental): Group C: Patients undergoing standard hepaticojejunostomy with no endoscopic access loop
  Interventions: Procedure: hepaticojejunostomy

INTERVENTIONS:
Procedure: hepaticojejunostomy — * Under general intubation anesthesia, a generous right subcostal incision is performed and could be extended on demand upward to the xiphoid process and/or to the left subcostal area. Thorough dissection and adhesiolysis is performed to reach the CBD and prepare the unaffected proximal part for anastomosis. The Roux jejunal loop is prepared and passed retrocolic to reach the porta hepatis.
  * Then, the hepaticojejunostomy is done via end to side anastomosis using interrupted sutures of polyglactin of 3-0 or 4-0 size. The anastomosis is done 10-15 cm away from the free distal end of the Roux jejunum loop to allow anastomosis without tension to the stomach. A biliary stent may be optionally placed according to operative circumstances and is brought out through the anterior abdominal wall.
  Arms: Group C:
Procedure: modified hepaticojejunostomy with subcutaneous access loop — In the subcutaneous access loop, the same steps are done for performing roux-en-Y hepaticojejunostomy.
  The closed free end of roux loop is passed through the anterior abdominal wall in the right subcostal area and then fixed to the wall in a subcutaneous position using 3/0 polyglactin sutures. The limb between the hepaticojejunal anastomosis and the subcutaneous fixation should be short and straight.
  Four Ligaclips are used to mark the jejunal loop by clipping the sutures holding the access loop in place.
  Arms: Group B:
Procedure: modified hepaticojejunostomy with gastric access loop — * In the gastric access loop, the same steps are done for performing roux-en-Y hepaticojejunostomy.The end of the Roux jejunal loop taken up for hepaticojejunostomy is not closed but is anastomosed to the anterior wall of the gastric antrum near the pyloric orifice.
  * All the enterogastrostomies and enteroenterostomies were in the form of single-layer continuous sutures of polyglactin of 3-0 size. An intraperitoneal drain was left in the hepatorenal pouch before closing the incision.
  Arms: Group A

SUMMARY:
Roux-en-Y hepaticojejunostomy is the standard procedure used by most hepatobiliary surgeons for biliary reconstruction following iatrogenic bile duct injury, benign and malignant CBD strictures, choledochal cysts and biliary tract tumors management. The incidence of anastomotic stricture following hepaticojejunostomy in experienced centers ranges between 5%-22%. Hepaticojejunostomy stricture is a serious complication of biliary surgery, if untreated, can lead to repeated cholangitis, intrahepatic stones formation, biliary cirrhosis, hepatic failure and eventually death.

Revision of hepaticojejunostomy is a complex procedure, the surgical procedure being made difficult by the sequelae of long-standing unrelieved biliary obstruction like portal hypertension due to secondary biliary cirrhosis, atrophy of liver lobes and presence of cholangiolytic liver abscess.

Endoscopic management is not only the least invasive but also very effective via either balloon dilatation or stenting of the stricture. In patients with "Roux-en-Y" hepaticojejunostomy, the endoscopic access to the anastomosis is hampered by the distance traveled by the jejunal loop until reaching the angle of the enteral anastomosis.

Many modifications of hepaticojejunostomy to provide permanent endoscopic access have been described in the literature including duodenal, gastric and subcutaneous access loops.

Gastric access loop was first described by Sitaram et al. Ten patients had undergone gastric access loop. Access loop was entered easily with the gastroscope in five patients in whom it was attempted. In a series with 16 cases, Hamad MA and El-Amin H assessed different construction of gastric access loop in the form of bilioenterogastrostomy the overall success rate of endoscopic access to the HJ through the three types of BEG was 87.5%, while it was 100% for BEG type III, which is a construction similar to the previous series (BEG) type.

Subcutaneous loop access was described by Chen et al. and by Huston et al. In Hutson's series of 7 patients, recurrent strictures were treated with repeated balloon dilations. The stone extractions were all successful. In most series, the subcutaneous loop was used for management os HJ stricture and intrahepatic stones by radiologic intervention. Recently the subcutaneous loop can be used as an endoscopic biliary access.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled study; which will include all patients who will undergo Roux-en-Y hepaticojejunostomy reconstruction during the period from 9-2017 to 12-2019.

* Methodology:

Patients will be randomized into three groups according to the surgical procedure performed as follows:

* Group A: Patients undergoing modified hepaticojejunostomy with gastric access loop
* Group B: Patients undergoing modified hepaticojejunostomy with subcutaneous access loop
* Group C: Patients undergoing standard hepaticojejunostomy with no endoscopic access loop

  * Pre-operative preparation:

For all patients, full medical history, clinical examination, laboratory investigations in the form of complete blood count (CBC), prothrombin time and concentration (PTT), liver function tests (LFT) and kidney function tests (KFT) will be performed.

Imaging studies will also be carried out in the form of abdominal ultrasonography (US), computerized tomography scan (CT) of the abdomen and magnetic resonance cholangiography (MRC) if indicated.

ERCP will be performed, whenever applicable, whether for diagnosis or therapeutic trial.

* Surgical Technique:

For gastric access loop:

* Surgical technique: under general intubation anesthesia, a generous right subcostal incision is performed and could be extended on demand upward to the xiphoid process and/or to the left subcostal area. Thorough dissection and adhesiolysis is performed to reach the CBD and prepare the unaffected proximal part for anastomosis. The Roux jejunal loop is prepared and passed retrocolic to reach the porta hepatis.
* Then, the hepaticojejunostomy is done via end to side anastomosis using interrupted sutures of polyglactin of 3-0 or 4-0 size. The anastomosis is done 10-15 cm away from the free distal end of the Roux jejunum loop to allow anastomosis without tension to the stomach. A biliary stent may be optionally placed according to operative circumstances and is brought out through the anterior abdominal wall.
* The end of the Roux jejunal loop taken up for hepaticojejunostomy is not closed but is anastomosed to the anterior wall of the gastric antrum near the pyloric orifice.
* All the enterogastrostomies and enteroenterostomies were in the form of single-layer continuous sutures of polyglactin of 3-0 size. An intraperitoneal drain was left in the hepatorenal pouch before closing the incision.

For subcutaneous access loop:

In the subcutaneous access loop, the same steps are done for performing roux-en-Y hepaticojejunostomy.

The closed free end of roux loop is passed through the anterior abdominal wall in the right subcostal area and then fixed to the wall in a subcutaneous position using 3/0 polyglactin sutures. The limb between the hepaticojejunal anastomosis and the subcutaneous fixation should be short and straight.

Four Ligaclips are used to mark the jejunal loop by clipping the sutures holding the access loop in place.

ELIGIBILITY:
Inclusion Criteria:

* All patients who will undergo roux-en-Y hepaticojejunostomy reconstruction at General surgery department - Assiut University.

Exclusion Criteria:

* Patients with malignant disease necessitating roux-en-Y hepaticojejunostomy (Cholangiocarcinoma or inoperable pancreatic cancer) will be excluded from this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
endoscopic access | first trial after 2 months (8 weeks) and second trial one year postoperatively
  two trial of endoscopic entry for assessment of hepaticojejunostomy after 2 months (8 weeks) and one year postoperatively

SECONDARY OUTCOMES:
mortality rate | up to 3 months postoperative for each case
  number of deaths intraoperative and postoperative related to surgery
bilio-enteric fistula | 1 month post-operative for each case, data will be available
  anastomotic leak from hepaticojejunostomy or enteroenterostomy
hepaticojejunostomy stricture | 6 months after the last case
  stricture at anastomotic site of hepaticojejunostomy that may occur at any time during the study and detected by development of obstructive jaundice If obstructive jaundice, biliary pain or cholangitis subsequently developed, abdominal ultrasonography followed by MRCP is then carried out. Thereafter, endoscopic assessment of the hepaticojejunostomy was done either by upper endoscopy in Group A or through skin incision and gastroendoscope or choledochoscope in Group B.
  Patients were reviewed 6 weeks after surgery, at 3-month intervals thereafter for the first year, and at 6-month intervals thereafter, unless they became symptomatic again.

IPD SHARING:
Plan to Share IPD: Undecided
All patients will be tested for liver functions tests and abdominal ultrasonography at the end of the 2nd post-operative week.
  All patients of Group A and B will undergo trial of endoscopic assessment after 2 months (8 weeks) and one year postoperatively.
  If obstructive jaundice, biliary pain or cholangitis subsequently developed, abdominal ultrasonography followed by MRCP is then carried out. Thereafter, endoscopic assessment of the hepaticojejunostomy was done either by upper endoscopy in Group A or through skin incision and gastroendoscope or choledochoscope in Group B.
  Patients were reviewed 6 weeks after surgery, at 3-month intervals thereafter for the first year, and at 6-month intervals thereafter, unless they became symptomatic again.

REFERENCES:
- [Background] Stewart L, Way LW. Bile duct injuries during laparoscopic cholecystectomy. Factors that influence the results of treatment. Arch Surg. 1995 Oct;130(10):1123-8; discussion 1129. doi: 10.1001/archsurg.1995.01430100101019. PMID 7575127
- [Background] Csendes A, Navarrete C, Burdiles P, Yarmuch J. Treatment of common bile duct injuries during laparoscopic cholecystectomy: endoscopic and surgical management. World J Surg. 2001 Oct;25(10):1346-51. doi: 10.1007/s00268-001-0121-5. PMID 11596901
- [Background] Davids PH, Tanka AK, Rauws EA, van Gulik TM, van Leeuwen DJ, de Wit LT, Verbeek PC, Huibregtse K, van der Heyde MN, Tytgat GN. Benign biliary strictures. Surgery or endoscopy? Ann Surg. 1993 Mar;217(3):237-43. doi: 10.1097/00000658-199303000-00004. PMID 8452402
- [Background] Alves A, Farges O, Nicolet J, Watrin T, Sauvanet A, Belghiti J. Incidence and consequence of an hepatic artery injury in patients with postcholecystectomy bile duct strictures. Ann Surg. 2003 Jul;238(1):93-6. doi: 10.1097/01.sla.0000074983.39297.c5. PMID 12832970
- [Background] Moraca RJ, Lee FT, Ryan JA Jr, Traverso LW. Long-term biliary function after reconstruction of major bile duct injuries with hepaticoduodenostomy or hepaticojejunostomy. Arch Surg. 2002 Aug;137(8):889-93; discussion 893-4. doi: 10.1001/archsurg.137.8.889. PMID 12146986
- [Background] Rothlin MA, Lopfe M, Schlumpf R, Largiader F. Long-term results of hepaticojejunostomy for benign lesions of the bile ducts. Am J Surg. 1998 Jan;175(1):22-6. doi: 10.1016/s0002-9610(97)00229-8. PMID 9445233
- [Background] Tocchi A, Costa G, Lepre L, Liotta G, Mazzoni G, Sita A. The long-term outcome of hepaticojejunostomy in the treatment of benign bile duct strictures. Ann Surg. 1996 Aug;224(2):162-7. doi: 10.1097/00000658-199608000-00008. PMID 8757379
- [Background] Lillemoe KD, Melton GB, Cameron JL, Pitt HA, Campbell KA, Talamini MA, Sauter PA, Coleman J, Yeo CJ. Postoperative bile duct strictures: management and outcome in the 1990s. Ann Surg. 2000 Sep;232(3):430-41. doi: 10.1097/00000658-200009000-00015. PMID 10973393
- [Derived] Raafat M, Morsy MM, Mohamed SI, Hamad MA, Sayed MM. Hepaticojejunostomy with gastric access loop versus conventional hepaticojejunostomy: a randomized trial. Updates Surg. 2023 Dec;75(8):2157-2167. doi: 10.1007/s13304-023-01604-6. Epub 2023 Aug 9. PMID 37556078